CLINICAL TRIAL: NCT02936999
Title: An Exploratory Pilot Study of Vitamin D Supplementation in Women With DCIS and/or LCIS
Brief Title: Vitamin D Supplementation in Women With DCIS and/or LCIS
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Terminated for lack of patient samples and funding
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-2399
Record Dates: First submitted 2016-10-11; First posted 2016-10-18 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vitamin D3 (Experimental): Patients will be dispensed cholecalciferol, 32 capsules/bottle of 1cap/4000 IU PO QD on Day 1 visit to take home. Bottle must be labeled with instructions on how to take the drug and the assigned patient ID number. Patients will be instructed to take 1 capsule per day, with water, for 29 days using the dispensed study bottle. They will be instructed to stop taking their daily vitamin D3 dose after 30 days of treatment. A study drug diary will be provided at Day 1 visit and patients will be instructed to complete the study drug diary daily from Day 2 to Day 30. Patient's report of vitamin-D3 intake from the diary must be reconciled against the number of capsules returned at Day 30 visit.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Cholecalciferol 100,000 IU followed by 4000 IU orally once daily for 30 days.
  Other Names: Vitamin D3

SUMMARY:
The purpose of this study is to determine the safety and usefulness of oral Vitamin D supplementation in subjects with in situ carcinoma. More specifically, this study is being done to (1) understand the effect of Vitamin D supplementation on behavior of breast cancer cells and (2) the development of invasive breast cancer disease.

DETAILED DESCRIPTION:
In vitro, calcitriol, the most potent metabolite of vitamin D, inhibits a variety of cellular pathways that promote cell proliferation and survival. Vitamin D has been shown to reduce the growth of breast cancer precursor cells in cell culture studies. In animal models Vitamin D has been shown to prevent the growth and progression of transplanted cell lines MCF710A, which is a model of pre-invasive cancer. Serum Vitamin D level deficiency correlates with an increased risk of breast cancer, and reduced survival of breast cancer patients. Vitamin D is also recognized to have effects on immune cell function and autoimmunity. The safety profile of oral Vitamin D, and its metabolite calcitriol, was well established for moderate term and acute therapy worldwide. Potential additional primary and secondary benefits of vitamin D are a) the suppression of carcinogen-induced transformation or progression of breast epithelium, and b) the enhancement of innate immune defense of pre-invasive breast cancer lesions, and c) its qualification as a combination therapy when combined with other neoadjuvant therapies for DCIS.

Patients who have been diagnosed by core biopsy with carcinoma in situ, ductal or lobular, will be evaluated for vitamin d supplementation. Patients with vitamin d levels less than 50 will be eligible for participation. They will receive a one month (30 days) schedule of vitamin D supplementation and then proceed with the standard of care of surgical excision. Immunohistochemistry studies will be performed on the diagnostic core biopsy and the surgical specimen to evaluate the impact of vitamin d supplementation on: the proliferative index-ki67, proliferative marker- PCNA, proteins of the autophagy pathway (LC3B, ATG7), her2 localization, and levels of PMCA2 - calcium efflux channel.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a tissue diagnosis of lobular carcinoma in situ or ductal carcinoma in situ and being scheduled to undergo excision of their cancer
* Subjects must be female at least 18 years of age
* Subjects must have a signed consent
* Normal liver function based on (total bilirubin and AST <1.5 x Upper Limit of Normal)
* Serum creatinine < 2.0 mg/dL
* Serum 25 (OH) D levels < 50 ng/ml
* Calcium within the normal range (8.5-10.2 mg/dL)
* ECOG performance status 0-2
* Are able to swallow and retain oral medication
* Subjects should be willing to abstain from use of hormonal therapies (e.g. hormone replacement therapy, oral contraceptive pills, hormone-containing IUDs, and E-string)

Exclusion Criteria:

* Patient desires not to participate in the study
* Inability to give consent
* Current use of hormone-containing forms of birth control such as implants (i.e. Norplants, or injectables (i.e. depo-provera)
* Currently lactating
* Patients with history of renal or hepatic insufficiency
* Used an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study medication
* History of granulomatous disease such as tuberculosis or sarcoidosis
* History of Vitamin D supplementation > 2000 IU/day within the last 2 months
* History of hypoparathyroidism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Wilkinson, MD, Principal Investigator — Inova Schar Cancer Institute
Locations (1):
- Inova Schar Cancer Institute, Fairfax, Virginia, United States

REFERENCES:
- [Background] Bernardes JR Jr, Nonogaki S, Seixas MT, Rodrigues de Lima G, Baracat EC, Gebrim LH. Effect of a half dose of tamoxifen on proliferative activity in normal breast tissue. Int J Gynaecol Obstet. 1999 Oct;67(1):33-8. doi: 10.1016/s0020-7292(99)00092-2. PMID 10576237
- [Background] Chen YY, DeVries S, Anderson J, Lessing J, Swain R, Chin K, Shim V, Esserman LJ, Waldman FM, Hwang ES. Pathologic and biologic response to preoperative endocrine therapy in patients with ER-positive ductal carcinoma in situ. BMC Cancer. 2009 Aug 18;9:285. doi: 10.1186/1471-2407-9-285. PMID 19689789
- [Background] Deeb KK, Trump DL, Johnson CS. Vitamin D signalling pathways in cancer: potential for anticancer therapeutics. Nat Rev Cancer. 2007 Sep;7(9):684-700. doi: 10.1038/nrc2196. PMID 17721433
- [Background] Espina V, Edmiston KH, Liotta LA. Non-enzymatic, serum-free tissue culture of pre-invasive breast lesions for spontaneous generation of mammospheres. J Vis Exp. 2014 Nov 8;(93):e51926. doi: 10.3791/51926. PMID 25406584
- [Background] Espina V, Liotta LA. What is the malignant nature of human ductal carcinoma in situ? Nat Rev Cancer. 2011 Jan;11(1):68-75. doi: 10.1038/nrc2950. Epub 2010 Dec 2. PMID 21150936
- [Background] Espina V, Mariani BD, Gallagher RI, Tran K, Banks S, Wiedemann J, Huryk H, Mueller C, Adamo L, Deng J, Petricoin EF, Pastore L, Zaman S, Menezes G, Mize J, Johal J, Edmiston K, Liotta LA. Malignant precursor cells pre-exist in human breast DCIS and require autophagy for survival. PLoS One. 2010 Apr 20;5(4):e10240. doi: 10.1371/journal.pone.0010240. PMID 20421921
- [Background] Esserman L. Neoadjuvant chemotherapy for primary breast cancer: lessons learned and opportunities to optimize therapy. Ann Surg Oncol. 2004 Jan;11(1 Suppl):3S-8S. doi: 10.1007/BF02524789. No abstract available. PMID 15015703
- [Background] Esserman L, Sepucha K, Ozanne E, Hwang ES. Applying the neoadjuvant paradigm to ductal carcinoma in situ. Ann Surg Oncol. 2004 Jan;11(1 Suppl):28S-36S. doi: 10.1007/BF02524793. PMID 15015707
- [Background] Fisher B, Costantino JP, Wickerham DL, Redmond CK, Kavanah M, Cronin WM, Vogel V, Robidoux A, Dimitrov N, Atkins J, Daly M, Wieand S, Tan-Chiu E, Ford L, Wolmark N. Tamoxifen for prevention of breast cancer: report of the National Surgical Adjuvant Breast and Bowel Project P-1 Study. J Natl Cancer Inst. 1998 Sep 16;90(18):1371-88. doi: 10.1093/jnci/90.18.1371. PMID 9747868
- [Background] Gandini S, Boniol M, Haukka J, Byrnes G, Cox B, Sneyd MJ, Mullie P, Autier P. Meta-analysis of observational studies of serum 25-hydroxyvitamin D levels and colorectal, breast and prostate cancer and colorectal adenoma. Int J Cancer. 2011 Mar 15;128(6):1414-24. doi: 10.1002/ijc.25439. PMID 20473927
- [Background] Gonzalez RJ, Buzdar AU, Fraser Symmans W, Yen TW, Broglio KR, Lucci A, Esteva FJ, Yin G, Kuerer HM. Novel clinical trial designs for treatment of ductal carcinoma in situ of the breast with trastuzumab (herceptin). Breast J. 2007 Jan-Feb;13(1):72-5. doi: 10.1111/j.1524-4741.2006.00366.x. PMID 17214797
- [Background] Hathcock JN, Shao A, Vieth R, Heaney R. Risk assessment for vitamin D. Am J Clin Nutr. 2007 Jan;85(1):6-18. doi: 10.1093/ajcn/85.1.6. PMID 17209171
- [Background] Alipour S, Hadji M, Hosseini L, Omranipour R, Saberi A, Seifollahi A, Bayani L, Shirzad N. Levels of serum 25-hydroxy-vitamin d in benign and malignant breast masses. Asian Pac J Cancer Prev. 2014;15(1):129-32. doi: 10.7314/apjcp.2014.15.1.129. PMID 24528013
- [Background] Hird RB, Chang A, Cimmino V, Diehl K, Sabel M, Kleer C, Helvie M, Schott A, Young J, Hayes D, Newman L. Impact of estrogen receptor expression and other clinicopathologic features on tamoxifen use in ductal carcinoma in situ. Cancer. 2006 May 15;106(10):2113-8. doi: 10.1002/cncr.21873. PMID 16596655
- [Background] Hwang ES, Esserman L. Neoadjuvant hormonal therapy for ductal carcinoma in situ: trial design and preliminary results. Ann Surg Oncol. 2004 Jan;11(1 Suppl):37S-43S. doi: 10.1007/BF02524794. PMID 15015708
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Jeong Y, Swami S, Krishnan AV, Williams JD, Martin S, Horst RL, Albertelli MA, Feldman BJ, Feldman D, Diehn M. Inhibition of Mouse Breast Tumor-Initiating Cells by Calcitriol and Dietary Vitamin D. Mol Cancer Ther. 2015 Aug;14(8):1951-61. doi: 10.1158/1535-7163.MCT-15-0066. Epub 2015 May 1. PMID 25934710
- [Background] Kaur P, Mishra SK, Mithal A. Vitamin D toxicity resulting from overzealous correction of vitamin D deficiency. Clin Endocrinol (Oxf). 2015 Sep;83(3):327-31. doi: 10.1111/cen.12836. Epub 2015 Jul 14. PMID 26053339
- [Background] Kumar AS, Bhatia V, Henderson IC. Overdiagnosis and overtreatment of breast cancer: rates of ductal carcinoma in situ: a US perspective. Breast Cancer Res. 2005;7(6):271-5. doi: 10.1186/bcr1346. Epub 2005 Nov 11. PMID 16457703
- [Background] Giammanco M, Di Majo D, La Guardia M, Aiello S, Crescimannno M, Flandina C, Tumminello FM, Leto G. Vitamin D in cancer chemoprevention. Pharm Biol. 2015;53(10):1399-434. doi: 10.3109/13880209.2014.988274. Epub 2015 Apr 9. PMID 25856702
- [Background] Lee O, Page K, Ivancic D, Helenowski I, Parini V, Sullivan ME, Margenthaler JA, Chatterton RT Jr, Jovanovic B, Dunn BK, Heckman-Stoddard BM, Foster K, Muzzio M, Shklovskaya J, Skripkauskas S, Kulesza P, Green D, Hansen NM, Bethke KP, Jeruss JS, Bergan R, Khan SA. A randomized phase II presurgical trial of transdermal 4-hydroxytamoxifen gel versus oral tamoxifen in women with ductal carcinoma in situ of the breast. Clin Cancer Res. 2014 Jul 15;20(14):3672-82. doi: 10.1158/1078-0432.CCR-13-3045. PMID 25028506
- [Background] Leonard GD, Swain SM. Ductal carcinoma in situ, complexities and challenges. J Natl Cancer Inst. 2004 Jun 16;96(12):906-20. doi: 10.1093/jnci/djh164. PMID 15199110
- [Background] Li CI, Malone KE, Saltzman BS, Daling JR. Risk of invasive breast carcinoma among women diagnosed with ductal carcinoma in situ and lobular carcinoma in situ, 1988-2001. Cancer. 2006 May 15;106(10):2104-12. doi: 10.1002/cncr.21864. PMID 16604564
- [Background] Li CI, Daling JR, Malone KE. Age-specific incidence rates of in situ breast carcinomas by histologic type, 1980 to 2001. Cancer Epidemiol Biomarkers Prev. 2005 Apr;14(4):1008-11. doi: 10.1158/1055-9965.EPI-04-0849. PMID 15824180
- [Background] Lopes N, Sousa B, Martins D, Gomes M, Vieira D, Veronese LA, Milanezi F, Paredes J, Costa JL, Schmitt F. Alterations in Vitamin D signalling and metabolic pathways in breast cancer progression: a study of VDR, CYP27B1 and CYP24A1 expression in benign and malignant breast lesions. BMC Cancer. 2010 Sep 11;10:483. doi: 10.1186/1471-2407-10-483. PMID 20831823
- [Background] Ma Y, Zhang P, Wang F, Yang J, Liu Z, Qin H. Association between vitamin D and risk of colorectal cancer: a systematic review of prospective studies. J Clin Oncol. 2011 Oct 1;29(28):3775-82. doi: 10.1200/JCO.2011.35.7566. Epub 2011 Aug 29. PMID 21876081
- [Background] Martin-Herranz A, Salinas-Hernandez P. Vitamin D supplementation review and recommendations for women diagnosed with breast or ovary cancer in the context of bone health and cancer prognosis/risk. Crit Rev Oncol Hematol. 2015 Oct;96(1):91-9. doi: 10.1016/j.critrevonc.2015.05.006. Epub 2015 May 19. PMID 26068240
- [Background] Pan H, Cai N, Li M, Liu GH, Izpisua Belmonte JC. Autophagic control of cell 'stemness'. EMBO Mol Med. 2013 Mar;5(3):327-31. doi: 10.1002/emmm.201201999. PMID 23495139
- [Background] Sanders KM, Stuart AL, Williamson EJ, Simpson JA, Kotowicz MA, Young D, Nicholson GC. Annual high-dose oral vitamin D and falls and fractures in older women: a randomized controlled trial. JAMA. 2010 May 12;303(18):1815-22. doi: 10.1001/jama.2010.594. PMID 20460620
- [Background] Schleck ML, Souberbielle JC, Jandrain B, Da Silva S, De Niet S, Vanderbist F, Scheen A, Cavalier E. A Randomized, Double-Blind, Parallel Study to Evaluate the Dose-Response of Three Different Vitamin D Treatment Schemes on the 25-Hydroxyvitamin D Serum Concentration in Patients with Vitamin D Deficiency. Nutrients. 2015 Jul 3;7(7):5413-22. doi: 10.3390/nu7075227. PMID 26151178
- [Background] Schnitt SJ. The transition from ductal carcinoma in situ to invasive breast cancer: the other side of the coin. Breast Cancer Res. 2009;11(1):101. doi: 10.1186/bcr2228. Epub 2009 Feb 27. PMID 19291276
- [Background] Wahler J, So JY, Kim YC, Liu F, Maehr H, Uskokovic M, Suh N. Inhibition of the transition of ductal carcinoma in situ to invasive ductal carcinoma by a Gemini vitamin D analog. Cancer Prev Res (Phila). 2014 Jun;7(6):617-26. doi: 10.1158/1940-6207.CAPR-13-0362. Epub 2014 Apr 1. PMID 24691501

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Patients will receive 100,000 IU PO loading dose at Day 1. The loading dose must be administered to the patient at the investigator's site.
Period: Overall Study
Arm/Group | Treatment Group
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Patients will receive 100,000IU PO loading dose at Day 1. The loading dose must be administered to the patient at the investigator's site.
Arm/Group | Treatment Group
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Ki 67 Measured
Description: The proliferation index measured by Ki67 will be described for both baseline (pre) and surgical (post) vitamin D supplementation. A paired t-test or the non-parametric Wilcoxon signed-rank test will be used when appropriate to compare patients' outcome between baseline and after-treatment.
Time Frame: 28 days +/- 3 days from Day 1 of treatment
Population: The study was terminated due to low enrollment and lack of funding; therefore no data were collected.
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

2. Secondary Outcome: Levels of Proteins of the Autophagy Pathway, LC3B
Description: Descriptive statistics (N, mean, median, Min, Max, STD for continuous variables, and N, proportion for categorical variables) will be used to summarize patients' demographics as well as lab results. . A paired t-test or the non-parametric Wilcoxon signed-rank test will be used when appropriate to compare patients' outcome between baseline and after-treatment. A p-value of <0.05 will be considered statistically significant.
Time Frame: 28 days +/- 3 days from Day 1 of treatment
Population: The study was terminated due to low enrollment and lack of funding therefore no data were collected.
Arm/Group | Vitamin D3
Number analyzed (Participants) | 0

3. Secondary Outcome: Levels of Proteins of the Autophagy Pathway, ATG7
Description: as for outcome 2
Time Frame: 28 days +/- 3 days from Day 1 of treatment
Population: The study was terminated due to low enrollment and lack of funding; therefore no data were collected.
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Levels of the Calcium Transport Proteins, PMCA2
Description: Descriptive statistics (N, mean, median, Min, Max, STD for continuous variables, and N, proportion for categorical variables) will be used to summarize patients' demographics as well as lab results. A paired t-test or the non-parametric Wilcoxon signed-rank test will be used when appropriate to compare patients' outcome between baseline and after-treatment. A p-value of <0.05 will be considered statistically significant.
Time Frame: 28 days +/- 3 days from Day 1 of treatment
Population: The study was terminated due to low enrollment and lack of funding; therefore no data were collected.
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

5. Secondary Outcome: HER2 Localization
Description: as for outcome 4
Time Frame: 28 days +/- 3 days from Day 1 of treatment
Population: The study was terminated due to low enrollment and lack of funding; therefore no data were collected.
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Clinical Assessment and adverse event evaluation will be done at Day 14, Day 21, and on the Post-Op visit on the study
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT02936999/Prot_SAP_000.pdf